CLINICAL TRIAL: NCT04685291
Title: Ultrasound-guided Block of the Supraclavicular Nerves for Clavicular Fractures in the Emergency Department
Brief Title: Ultrasound-guided Block of the Supraclavicular Nerves in Clavicular Fractures
Acronym: US-SCNB_Clav
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eckehart SCHÖLL (Other)
Responsible Party: Sponsor-Investigator, Eckehart SCHÖLL, Head of Emergency Department, Merian Iselin Klinik
Organization: Merian Iselin Klinik (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.0 / 10.12.2020
Record Dates: First submitted 2020-12-14; First posted 2020-12-28 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Clavicular Fracture; Pain, Acute
Keywords: ultrasound-guided regional anesthesia; Clavicular fracture; Emergency Department; pain management
MeSH Terms: conditions — Acute Pain; Emergencies; Agnosia

STUDY DESIGN:
Intervention Model Description: Prospective randomised single centre study
Masking Description: The comparator group will get systemic conventional pain management. Pain management using placebo would be harmful in patients with clavicular fractures. If these patients will have a severely dislocated fracture, they will be scheduled to have internal fixation of the fracture within the next 24 hours. They will receive oral and intravenous pain management.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Control (Active Comparator): Systemic conventional pain management. Adult patients with acute fractures of the clavicle, who are scheduled to have internal fixation of the fracture within the next 24 hours receive oral and intravenous pain management.
  Interventions: Drug: Conventional pain management
- Group 2: Nerve Block (Active Comparator): Adult patients with acute fractures of the clavicle, who are scheduled for an internal fixation of the fracture within the next 24 hours will receive an ultrasound-guided block of the supraclavicular nerves using a maximum of 3 ml of a long-acting local anesthetic. The injection is carried out directly in the emergency department following a sonographic or radiological diagnosis.
  Interventions: Procedure: Ultrasound-guided block of the supraclavicular nerves

INTERVENTIONS:
Procedure: Ultrasound-guided block of the supraclavicular nerves — The supraclavicular nerves (SCN) arise from the 3rd and 4th roots of the spinal nerves. After emerging from the spine, they run at the rear margin of the sternocleidomastoid muscle and divide into their three terminal branches. With a high-resolution Ultrasound (US)-probe they can be visualized as a grape-like structure under the skin. At this location, patient's skin is disinfected and covered with a sterile perforated blanket. The US-probe is covered with a sterile sheath. The patient is positioned as comfortably as possible so that the broken clavicle is not mobilized. SCN are shown by US and a 0.5 mm needle is advanced through the patient's skin in order to direct it to the nerves under US-guidance. Both the nerves and the needle are permanently visualized. As soon as the needle tip is placed next to the SCN, 2-3 millilitres of a long-acting LA are injected. The distribution of the LA around the nerves is controlled.
  Arms: Group 2: Nerve Block
Drug: Conventional pain management — * oral pain medication in patients younger than 70 years: Ibuprofen 400mg (1-1-1) AND Metamizole 500mg (max. 2 tbl. every 6 hours)
  * oral pain medication in patients older than or equal 70 years: Acemetacin 60mg (1-1-1) AND Metamizole 500mg (max. 2 tbl. every 6 hours)
  * Rescue analgesic medication for all patients: oxycodone hydrochlorid (drops) p.o. (10 mg/ml) 0.1mg/kg p.o. hour
  * In the ED Rescue analgesic medication for all patients: Fentanyl 50mcg i.v. (max. 200mcg/hour)
  Arms: Group 1: Control

SUMMARY:
A Clavicular fractures (CF) is uncomfortable for the affected patients because the fragments are often strongly displaced by the muscles attached to them and the bony fragments move painfully with every movement of the shoulder. In emergency departments (ED), so far CF has been tackled with drugs that are taken by mouth or injected into a vein. This type of pain management has many side effects since these painkillers act systemically.

The aim of the study is to investigate the effectiveness of pain relief in CF to be operated using regional anaesthesia. For this purpose, the supraclavicular nerves (SCN), which run directly under the skin of the neck, will be located using an ultrasound device (US). Under US-guidance the injection needle approaches the SCN and 2-3 millilitres of local aesthetic (LA) are injected around the nerves. The pain relief may last 12 up to 24 hours, which bridges the time until the operation (OP).

In order to compare this procedure, CF-patients will be divided into two groups, of which the control group (21) will be treated with painkillers in the conventional manner and the intervention group (21) will receive the US-guided block of the SCN.

With the small amount of LA injected, adverse events (AE) are very rare. Nevertheless, the puncture in the side of the neck may cause bruises at the site of the injection or uncomfortable, spreading pain. Systemic side effects are unlikely.

In the intervention group, the investigators expect a nearly complete pain relief up to the operation than with conventional pain therapy and a lower rate of side effects than with systemic administration of painkillers.

DETAILED DESCRIPTION:
In 2013 Tran and colleagues reported about a controversial knowledge concerning the sensory innervation of the clavicle which may lead to different approaches of regional analgesia (RA) in CF: superficial cervical plexus blocks, interscalene blocks, and combined superficial cervical plexus-interscalene blocks. Since the innervation of the clavicle comes from four nerves (supraclavicular nerves, subclavian nerve, long thoracic nerve and suprascapular nerve) it seams to be quite difficult to guarantee a complete sensible clavicular block for an operation. Nevertheless, few case reports exist, witch describe clavicle operations under RA alone. However, in these cases a considerable amount of local anaesthetics (LA) has been used that it may be assumed that there could have been dangerous side effects.

Valdés-Vilches and Sánchez-del Águila pronounced the importance of the supraclavicular nerves (SCN) in CF. For that reason, our purpose is to determine the effectivity of a single nerve block of SCN in CF in the ED with only 2-3 millilitres of LA. The aim of our study is to investigate the effectiveness of this method in CF to be operated up to 24 hours later. For this purpose, the SCN, which run directly under the skin of the neck, will be located using an ultrasound device (US). Under US-guidance the injection needle approaches the SCN and 2-3 millilitres of LA are injected around the nerves. The pain relief may last 12 up to 24 hours, which bridges the time until the operation (OP).

In order to compare this new procedure, CF-patients will be divided into two groups, of which the control group (20) will be treated with painkillers in the conventional manner and the intervention group (20) will receive the US-guided block of the SCN.

The following medical products and medicaments will be used, which are all already registered and authorised in Switzerland:

* US-machines: Samsung HS60 High-End with linear-probe (array) LA4-18BD; Samsung RS85 Premium Radiology with linear probe LA4-18B.
* Needle: PAJUNK SonoTAP 24 Gauge x 40mm
* LA: 3 ml Bupivacaine 0.5% +75mcg Clonidine as an adjuvant. The LA will be used in accordance with the prescribing information. The dose will be up to 10 fold lower than the usual used dosages in cervical nerve blocks, since with US-guidance there will be an excellent accuracy to approach the desired single nerve.

In the intervention group, the investigators expect a nearly complete pain relief up to the operation than with conventional pain management and a lower rate of side effects than with systemic administration of painkillers.

With the small amount of LA injected, adverse events (AE) are expected very rare. Nevertheless, the puncture in the side of the neck may cause bruises at the site of the injection or uncomfortable, spreading pain. Systemic side effects are unlikely. A well-known and much feared AE of RA of the brachial and cervical plexus is accidental anaesthesia of the phrenic nerve, which runs from the neck to the diaphragm near the four aforementioned nerves. The paralysis of the phrenic nerve by the injected LA can cause breathing difficulties because the diaphragm is the main breathing muscle. Another possible complication is a drop in blood pressure and heart rate, which can result from anaesthesia of the autonomic nerves in the neck. For these reasons, RA of the brachial and cervical plexus should be performed with as little LA as possible. However, if the SCN-block is performed correctly, the LA can neither reach the phrenic nerve nor the vegetative nerves, since the SCN lays outside the prevertebral layer of the deep cervical fascia, where the phrenic and the vegetative nerves lie within.

Preliminary investigations in our ED in the last two years have shown that 2-3 millilitres of LA are too small a quantity of fluid to reach the phrenic nerve or to cause serious systemic side effects through absorption.

ELIGIBILITY:
Inclusion Criteria:

* adult ED-patients with sonographic and / or radiologically diagnosed clavicular fracture, who are scheduled for operation within the next 24 hours
* older then 18 years
* no known allergies to local anesthetic drugs

Exclusion Criteria:

* refusal of the procedure by the patient
* infection at the site of possible injection of local anaesthetics
* known allergies against local anaesthetics
* inability of consent or no carer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | within the first 24 hours after ED-Admission or until the operation
  The numerical rating scale (NRS) is one of the most widely used pain rating scales. It ranges from zero to ten, with zero being no pain and ten being the worst possible pain. The measurement of the NRS is achieved using the patient evaluation sheet.

SECONDARY OUTCOMES:
Painkillers in milligrams until surgery | within the first 24 hours after ED-Admission or until the operation
  The painkillers that are required before the operation or within the first 24 hours are listed and divided into the various classes of action. The respective amounts will be given in milligrams.
Painkillers in milligrams after surgery | within the first 24 hours after ED-Admission after the operation
  The painkillers that are required after the operation within 24 hours are listed and divided into the various classes of action. The respective amounts will be given in milligrams.
Patient Questionnaire | Within the first 24 hours after ED-Admission or after operation
  After 24 hours the patients of both groups will be given a questionnaire with the following questions:
  1. Were you satisfied with the overall pain management?
     Possible answers:
     * not at all
     * less
     * fair
     * good
     * excellent
  2. Did you have any pain in the first 24 hours?
     Possible answers:
     * extreme
     * severe
     * moderate
     * less
     * no pain
  3. For block patients only: How did you experience the procedure?
     Possible answers:
     * very unpleasant
     * unpleasant
     * ok
     * good
     * excellent
  4. Were you satisfied with the pain management on the ED?
     Possible answers:
     * dissatisfied
     * less satisfied
     * ok
     * good
     * excellent
  5. For block patients only: Would you have the block done again?
  Possible answers:
  * no
  * rather not
  * don't know
  * probably
  * yes
Incidence of side effects | within the first 24 hours after ED-Admission
  The incidence of side effects in both groups:
  * neuralgic pain due to the puncture
  * bruise at the point of LA-injection
  * infection at the site of the puncture
  * breathing difficulties: accidental anaesthesia of the phrenic nerve
  * accidental anaesthesia of other nerves of the cervical plexus
  * prolonged drop in blood pressure and heart rate: accidental anaesthesia of the sympathetic nervous system

CONTACTS AND LOCATIONS:
Overall Officials: Eckehart Schöll, MD, Principal Investigator — Merian Iselin Klinik
Locations (1):
- Merian Iselin Klinik, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared with other researchers.

REFERENCES:
- [Background] Tran DQ, Tiyaprasertkul W, Gonzalez AP. Analgesia for clavicular fracture and surgery: a call for evidence. Reg Anesth Pain Med. 2013 Nov-Dec;38(6):539-43. doi: 10.1097/AAP.0000000000000012. PMID 24121609
- [Background] Shanthanna H. Ultrasound guided selective cervical nerve root block and superficial cervical plexus block for surgeries on the clavicle. Indian J Anaesth. 2014 May;58(3):327-9. doi: 10.4103/0019-5049.135050. PMID 25024480
- [Background] Ueshima H, Otake H. Successful clavicle fracture surgery performed under selective supraclavicular nerve block using the new subclavian approach. JA Clin Rep. 2016;2(1):34. doi: 10.1186/s40981-016-0061-6. Epub 2016 Nov 8. PMID 29492429 (Retraction: PMID 32494982 JA Clin Rep. 2020 Jun 3;6(1):40)
- [Background] Valdes-Vilches LF, Sanchez-del Aguila MJ. Anesthesia for clavicular fracture: selective supraclavicular nerve block is the key. Reg Anesth Pain Med. 2014 May-Jun;39(3):258-9. doi: 10.1097/AAP.0000000000000057. No abstract available. PMID 24747317
- [Background] Popping DM, Elia N, Marret E, Wenk M, Tramer MR. Clonidine as an adjuvant to local anesthetics for peripheral nerve and plexus blocks: a meta-analysis of randomized trials. Anesthesiology. 2009 Aug;111(2):406-15. doi: 10.1097/ALN.0b013e3181aae897. PMID 19602964
- [Background] Wadlund DL. Local Anesthetic Systemic Toxicity. AORN J. 2017 Nov;106(5):367-377. doi: 10.1016/j.aorn.2017.08.015. PMID 29107256